CLINICAL TRIAL: NCT02643667
Title: A Phase 2 Study of Ibrutinib as Neoadjuvant Therapy in Patients With Localized Prostate Cancer
Brief Title: Ibrutinib as Neoadjuvant Therapy in Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201808057
Record Dates: First submitted 2015-12-28; First posted 2015-12-31 (Estimated); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: Radical prostatectomy (RP)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I: Ibrutinib (Experimental): * Ibrutinib 840 mg by mouth once daily for 2 weeks.
  * Radical prostatectomy will be performed at least 7 days but not more than 12 days following the last scheduled dose of ibrutinib.
  Interventions: Drug: Ibrutinib; Procedure: Radical prostatectomy
- Safety Run-In and Phase II: Ibrutinib (Experimental): * Ibrutinib 840 mg by mouth once daily for 4 weeks.
  * Radical prostatectomy will be performed at least 7 days but not more than 12 days following the last scheduled dose of ibrutinib
  Interventions: Drug: Ibrutinib; Procedure: Radical prostatectomy

INTERVENTIONS:
Drug: Ibrutinib — -Ibrutinib will be supplied by Pharmacyclics Inc.
Procedure: Radical prostatectomy — -Standard of care

SUMMARY:
30-40% of patients who undergo radical prostatetecomy (RP) with curative intent for their localized prostate cancer experience relapse of their disease. Thus, improved therapeutic approaches are needed in this patient population. Enhancing the patient's anti-tumor immune response prior to surgery may improve long-term outcomes following RP

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* ECOG performance status 0 or 1
* Histologically documented adenocarcinoma of the prostate
* Patients must be suitable for and willing to undergo a radical prostatectomy at the completion of study therapy.
* Adequate bone marrow function, defined as:

  * WBC >2,500 cells/mm3
  * ANC >1,500 cells/mm3
  * Hemoglobin >9 mg/dL
  * Platelet count >100,000 cells/mm3
* Adequate renal function, defined as serum creatinine <2 mg/dL or CrCl >30 mL/min
* Adequate liver function, defined as:

  * AST and ALT <2.5x institutional ULN
  * Serum bilirubin <1.5x institutional ULN
* Adequate coagulation function, defined as normal PT/INR and PTT
* Ability to understand and willingness to sign a written informed consent document
* Available evaluable archival tumor tissue for correlative studies including assessment of immune infiltration and Btk expression is required. If archival tissue is unavailable, patients must be willing to undergo repeat prostate biopsy. Tissue is considered sufficient for correlative endpoint analyses if they are obtained from at least 2 prostate cores and consist of at least 15 unstained slides from the largest tumor volume and/or highest Gleason score. The availability of archival tissue or consent for repeat prostate biopsy is required for study eligibility; determination of tissue sufficiency is not required for study eligibility.
* The effects of ibrutinib on the developing human fetus is unknown. Men treated or enrolled on this protocol must agree to use adequate contraception prior to the study, for the duration of the study participation, and for 3 months after completion of treatment.

Exclusion Criteria:

* Patients with neuroendocrine or small cell features are not eligible.
* Any evidence of metastatic disease. Pre-operative staging will be undertaken per urologic standard of care.
* Any prior use of hormonal therapy, including:

  * GNRH agonists or GNRH antagonists (e.g., leuprorelin, degarelix)
  * Antiandrogens (e.g., bicalutamide, flutamide, nilutamide)
  * Novel androgen-directed therapies (e.g., abiraterone, enzalutamide)
  * Any estrogen containing compounds
  * 5-alpha reductase inhibitors (e.g., finasteride, dutasteride)
  * PC-SPES or PC-x products. Other herbal therapies or supplements will be considered by the Principle Investigator on a case by case basis based on their potential for hormonal or anti-cancer therapies.
* Chemotherapy ≤ 21 days prior to first administration of study treatment and/or monoclonal antibody ≤ 6 weeks prior to first administration of study treatment
* Prior radiation therapy for prostate cancer
* Prior exposure to BTK inhibitors
* Prior investigational therapy for prostate cancer
* Patients may not receive any other concurrent investigational agents while on study.
* Use of systemic steroid therapy within 28 days of study screening. Patients on inhaled or topical steroids are eligible.
* Concurrent systemic immunosuppressive therapy within 21 days of the first dose of study drug.
* Major surgery requiring the use of general anesthetic within 4 weeks of study enrollment
* HIV, active hepatitis B (HBV) or active hepatitis C (HCV)

  * Patients with past HBV infection or resolved HBV infection, defined as the presence of hepatitis B core antibody (HBc Ab) and absence of hepatitis B surface antigen (HBsAg) are eligible. HBV DNA must be obtained in these patients prior to day 1 of ibrutinib therapy, but detection of HBV DNA in these patients will not exclude study participation.
  * Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Inability to swallow capsules or presence of malabsorption syndromes, disease significantly affecting gastrointestinal function, history of resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete small obstruction.
* Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Function Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to screening.
* Uncontrolled concurrent illness, or any underlying medical condition, which in the Principal Investigator's opinion will make the administration of ibrutinib hazardous or obscure the interpretation of adverse events.
* Recent infection requiring systemic treatment that was completed within 14 days prior to the first dose of study drug
* Concurrent active malignancy other than non-melanoma skin cancers. Patients are considered to be free of active malignancy if they have completed curative therapy and have a <30% risk of relapse.
* History of congenital bleeding diathesis.
* Known bleeding disorders (e.g. von Willebrand's disease or hemophilia).
* Concomitant use of anticoagulants including warfarin, other Vitamin K antagonists, and enoxaparin.
* Subjects who received a strong or moderate cytochrome P450 (CYP) 3A4 inhibitor within 7 days prior to the first dose of ibrutinib or patients who require treatment with a strong or moderate cytochrome P450 (CYP) 3A inhibitor.
* Vaccination with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Patients on anti-platelet agents including clopidogrel and glycoprotein IIb/IIIa inhibitors. Aspirin is allowed, but should be held before surgery according to standard practices.
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child-Pugh classification
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to CTCAE v 4.03 grade 0 or 1 or to the levels dictated in the eligibility criteria with the exception of alopecia.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell K Pachynski, M.D., Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase I: Ibrutinib | Safety Run-In and Phase II: Ibrutinib
Started | 3 | 24
Completed | 3 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Ibrutinib | Safety Run-In and Phase II: Ibrutinib | Total
Number analyzed (Participants) | 3 | 24 | 27
Age, Continuous [Median (Full Range); unit: years] | 61 [56 to 67] | 62.5 [45 to 74] | 61 [45 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 24 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 24 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 24 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 24 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (Phase I and Safety Run-In)
Description: * CTCAE v.4.0
  * DLTs will be defined as any of the following that are attributable to ibrutinib.
    * Any grade 4 toxicity, including hematologic toxicities with the exception of lymphocytosis. Lymphocytosis, in the absence of clinical symptoms, is excluded from DLT, as this may be considered an on-target pharmacodynamics effect of BTK inhibition.
    * Any grade 3 toxicity.
    * Any recurrence of the same grade 3 toxicity.
    * Any delay of RP due to study-drug related toxicity.
    * Any complications of RP (e.g., bleeding, delayed wound healing) deemed to be related to study drug.
Time Frame: Completion of DLT follow-up (2 weeks for Phase I portion and 28 days for Safety Run-In)
Population: Only participants enrolled in the Phase I portion and the 6 participants in the Safety Run-In portion of the Phase II portion are evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ibrutinib | Safety Run-In and Phase II: Ibrutinib
Number analyzed (Participants) | 3 | 6
Participants | 0 | 0

2. Primary Outcome: Percentage of Participants With Positive Responses - CD20+ B Cells, IL-10+ B Cells, CD3+ T Cells, CD8+ Cytotoxic T Cells, Effector CD4+FOXP3- T Cells, and CD4+FOX3+ T Regulatory Cells
Description: In pre-treatment biopsy, RP tissue, and reference RP tissue quantitated by immunohistochemistry (IHC). Patients will be considered to have a positive response if there is >2 fold decrease from pre-treatment to post-treatment, or considered to have a negative response if there is <2 fold decrease. The percentage of participants who have "positive" responses are represented in the outcome measure data.
Time Frame: Pre-treatment and at time of RP (approximately 10 weeks after start of treatment)
Population: Only those in the Safety Run-In and Phase II portion were evaluable for this outcome measure. Additional participants in the Safety Run-In were not analyzed for this outcome measure due to either missing sample or too few cells in the sample to analyze. The investigators were unable to analyze matched/paired samples due to sample processing issues with the enrolled patients diagnostic biopsies (not enough evaluable tissue or unable to obtain biopsy tissue from outside medical center).
Measure: Number; unit: percentage of participants
Arm/Group | Phase I: Ibrutinib | Safety Run-In and Phase II: Ibrutinib
Number analyzed (Participants) | 0 | 15
percentage of participants
  CD20+ B cells: number analyzed (Participants) | 0 | 13
  CD20+ B cells |  | 53.8
  IL10+ B cells |  | 40
  CD3+ T cells: number analyzed (Participants) | 0 | 14
  CD3+ T cells |  | 7.1
  CD8+ T cells |  | 0
  CD4+ Foxp3- T cells |  | 0
  CD4+ Foxp3+ T cells |  | 13.3

3. Primary Outcome: Mean B Cell Fold Change of CD20+ B Cells
Description: Participants will be considered to have a positive response if there is >2 fold decrease (0.5 or less B cell fold change) or considered to have a negative response if there is <2 fold decrease. Descriptive statistics will be used to describe pre-treatment biopsy immune infiltration, post-treatment RP immune infiltration, and immune infiltration of reference RP tissue.
Time Frame: At RP (approximately 10 weeks after start of treatment)
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: B cell fold change
Groups:
- Phase I: Ibrutinib: * Ibrutinib 840 mg by mouth once daily for 2 weeks.
  * Radical prostatectomy will be performed at least 7 days but not more than 12 days following the last scheduled dose of ibrutinib.
  I
Arm/Group | Phase I: Ibrutinib | Safety Run-In and Phase II: Ibrutinib
Number analyzed (Participants) | 0 | 13
B cell fold change |  | 0.9 [0.3 to 1.5]

4. Secondary Outcome: Percentage of Participants With Positive Responses - CD19+ B Cells, CD25^highCD27^highCD86^High B Regulatory Cells, and CD3+, CD8+, CD4+FOXP3- and CD4+FOXP3+ T Cells Induced by Neoadjuvant Ibrutinib in Patients by Flow Cytometry
Description: Patients will be considered to have a positive response if there is >2 fold decrease from pre-treatment to post-treatment, or considered to have a negative response if there is <2 fold decrease. The percentage of partcipants who have "positive" responses are represented in the outcome measure data.
Time Frame: Pre-treatment to RP (approximately 10 weeks after start of treatment)
Population: Only those in the Safety Run-In and Phase II portion were evaluable for this outcome measure. Additional participants in the Safety Run-In were not analyzed for this outcome measure due to either missing sample or too few cells in the sample to analyze.
Measure: Number; unit: percentage of participants
Arm/Group | Phase I: Ibrutinib | Safety Run-In and Phase II: Ibrutinib
Number analyzed (Participants) | 0 | 21
percentage of participants
  CD19+ B cells |  | 38.1
  CD25+CD27+CD86+ regulatory B cells: number analyzed (Participants) | 0 | 20
  CD25+CD27+CD86+ regulatory B cells |  | 35
  CD3+ T cells |  | 14.3
  CD8+ T cells |  | 9.5
  CD4+ Foxp3- T cells |  | 14.3
  CD4+ Foxp3+ T cells |  | 14.3

5. Secondary Outcome: Number of Participants Who Had a 50% or Greater Decline in PSA
Time Frame: At baseline and approximately day 29
Population: If participants did not have the day 29 PSA drawn then they are not included in the overall number of participants analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ibrutinib | Safety Run-In and Phase II: Ibrutinib
Number analyzed (Participants) | 3 | 23
Participants | 0 | 0

6. Secondary Outcome: Number of Participants With a Treatment Response (Safety Lead-In and Phase II Only)
Description: Pathologic down-staging and/or pathologic T0
Time Frame: Completion of follow-up (approximately 10 weeks after start of treatment)
Population: Only participants in the Safety Lead-In and Phase II portion of the study who had a radical RP are evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: Ibrutinib | Safety Run-In and Phase II: Ibrutinib
Number analyzed (Participants) | 0 | 21
Participants |  | 7

ADVERSE EVENTS:
Time Frame: - Adverse events were collected from start of treatment until 30 days after the end of treatment (up to a total of 6 weeks for Phase I portion and up to 2 months for Safety Run-In and Phase II portion). - All-cause mortality was collected from start of treatment until completion of follow-up (up to week 10, approximately day 64).
Arm/Group | Phase I: Ibrutinib | Safety Run-In and Phase II: Ibrutinib
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/3 | 5/24
Other Adverse Events (participants affected / at risk) | 3/3 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Ibrutinib (N=3) | Safety Run-In and Phase II: Ibrutinib (N=24)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Fever (General disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Lymphocele (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: Ibrutinib (N=3) | Safety Run-In and Phase II: Ibrutinib (N=24)
Anemia (Blood and lymphatic system disorders) | 0 | 15
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3
Bilateral ear aches (Ear and labyrinth disorders) | 0 | 1
Right peripheral vision loss (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 10
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Flatulence (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 7
Stomach pain (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 3
Tongue wound (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Chest tightness (General disorders) | 0 | 1
Chills (General disorders) | 0 | 2
Edema (General disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 11
Fever (General disorders) | 0 | 1
Generalized body aches (General disorders) | 0 | 1
Lip swelling (General disorders) | 0 | 1
Pain (General disorders) | 2 | 1
Sweating (General disorders) | 0 | 1
Possible post-surgical infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Brusing (Injury, poisoning and procedural complications) | 0 | 1
Sore at incision site (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 5
Alkaline phosphatase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 4
Creatinine increased (Investigations) | 0 | 7
Lymphocyte count decreased (Investigations) | 0 | 1
Lymphocyte count increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 5
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain of bilateral Achilles tendon (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 5
Headache (Nervous system disorders) | 0 | 6
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 3
Hematuria (Renal and urinary disorders) | 0 | 3
Proteinuria (Renal and urinary disorders) | 0 | 4
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 1
Sharp pain in prostate (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus drainage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Blistering rash on hand (Skin and subcutaneous tissue disorders) | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritic rash (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash NOS (Skin and subcutaneous tissue disorders) | 0 | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4
Rash/bumps on scalp (Skin and subcutaneous tissue disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Lymphedema (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT02643667/Prot_SAP_000.pdf